CLINICAL TRIAL: NCT06762015
Title: Practice Environment for Nursing and Patient Safety in Primary Health Care
Brief Title: Nursing Practice Environment and Patient Safety in Primary Health Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cintia Silva Fassarella (Other)
Collaborators: CINTESIS - Center for Health Technology and Services Research, Porto (Unknown); Universidade do Porto (Other)
Responsible Party: Sponsor-Investigator, Cintia Silva Fassarella, Professor Dr., Rio de Janeiro State University
Organization: Rio de Janeiro State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CES n. 57_2024
Record Dates: First submitted 2024-12-26; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Healthy Work Environment; Patient Safety; Primary Health Care
Keywords: Healthy Work Environment; Patient Safety; Primary Health Care; Nurses

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Stratified random sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who will undertake the Positive Nursing Practice Environments Promotion Program
  Interventions: Behavioral: Positive Nursing Practice Environments Promotion Program
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Positive Nursing Practice Environments Promotion Program — A multi-component intervention program aimed at promoting positive nursing practice environments.
  Arms: Intervention Group

SUMMARY:
The goal of this study is to conduct an experimental, controlled, and randomized study, which will involve two data collection points - pre-intervention, post-intervention and a follow-up to asses the impact of the program. The study will be carried out with two groups - an intervention group and a control group, consisting of nurses interested in participating in the Positive Nursing Practice Environments Promotion Program (PAPEP), a multi-component intervention program aimed at promoting positive nursing practice environments. Participant allocation will be conducted randomly, using software to ensure stratified randomization of participants between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in primary health care units

Exclusion Criteria:

* Nurses in primary health care who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Work Environment | 6 months
  Scale for the environments evaluation of professional nursing practice-shortened version.
  The Scale for the Environment's Evaluation of Professional Nursing Practice-Shortened Version consists of 59 items across three subscales: Structure (29 items), Process (19 items), and Outcome (11 items). Participants rate each item on a five-point Likert scale (1: never to 5: always). Higher scores indicate a more favorable nursing practice environment for care quality and professional well-being. Scores are interpreted as follows: <35% (unfavorable), 35-55% (moderately favorable), 55-75% (favorable), and >75% (very favorable).
Safety climate | 6 months
  Safety Attitudes Questionnaire - Short Form The Safety Attitudes Questionnaire (SAQ) - Short Form 2006 assesses healthcare professionals' perceptions of patient safety attitudes across various clinical areas and healthcare services. It has been validated and culturally adapted to the context in which the study will be conducted. The SAQ - Short Form 2006 comprises six dimensions, addressing organizational factors, work environment factors, and team factors, with a total of 30 items. Participants respond to each item using a five-point Likert scale: "strongly disagree," "partially disagree," "neutral," "partially agree," and "strongly agree." The final score ranges from 0 to 100, where 0 represents the worst perception and 100 the best perception of the safety climate.

CONTACTS AND LOCATIONS:
Locations (1):
- ULS Entre Douro e Vouga, Santa Maria da Feira, Aveiro District, Portugal